CLINICAL TRIAL: NCT00303979
Title: Registry to Improve the Use of Evidence-Based Heart Failure Therapies in the Outpatient Setting
Brief Title: IMPROVE HF: Registry to Improve the Use of Evidence-Based Heart Failure Therapies in the Outpatient Setting
Acronym: IMPROVE-HF
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 258
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure, Congestive; Myocardial Infarction; Ventricular Dysfunction, Left
Keywords: Systolic Heart Failure; Quality of Care; Outcomes; Evidence-based Guidelines; Recommended Therapies
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Ventricular Dysfunction, Left; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort A (longitudinal): Longitudinal Cohort: Approximately 15,000 patients followed at baseline, 12 months and 24 months
- Cohort B (6 Month): 6 Month Cohort: Approximately 10,000 patients reviewed at single time point
- Cohort C (18 Month): 18 Month Cohort: Approximately 10,000 patients reviewed at single time point

SUMMARY:
The purpose of this study is to characterize current management of patients with either heart failure or prior myocardial infarction and left ventricular dysfunction and to assess the effect of education, specific clinical guidelines, reminder systems, comprehensive disease state management tools, benchmarked quality reports, and academic detailing on the use of evidence-based heart failure therapies in cardiology practices. This study is a quality improvement initiative that is being conducted through review of patient records.

DETAILED DESCRIPTION:
IMPROVE HF, the largest US outpatient HF patient registry, has substantially contributed to our knowledge of how systolic HF and post MI left ventricular systolic dysfunction (LVSD) patients are treated in the outpatient setting.

The findings of IMPROVE HF clearly support this guideline and may help to establish a model framework for future performance improvement programs for outpatient cardiology practices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Primary or secondary diagnosis of heart failure or prior myocardial infarction (heart attack)
* Moderate-to-severe left ventricular dysfunction (LVD) as demonstrated by an ejection fraction < or = 35% and/or a qualitative assessment of LVD of moderate-to-severe or severe LVD
* Patient has been seen at the clinic at least twice in the past 2 years
* Patient received care from the physician participating in the study

Exclusion Criteria:

* Patient has died
* Patient is not expected to survive for 12 months due to medical conditions other than heart failure
* Patient has undergone heart transplant surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients in outpatient cardiology practices
Sampling Method: Probability Sample
Enrollment: 34810 (Actual)
Dates: Start 2005-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Fonarow, MD, Study Chair — University of California at Los Angeles; Clyde Yancy, MD, Study Chair — UT Southwestern Medical Center at Dallas
Locations (141):
- United States (141):
  - Cardiovascular Associates of Montclair, Birmingham, Alabama
  - Cardiology Associates, Mobile, Alabama
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Heart Care, PC, Scottsdale, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Central Arkansas Cardiovascular Institute, Hot Springs, Arkansas
  - Arkansas Cardiology Clinic, Little Rock, Arkansas
  - St. Jude Heritage Medical Group, Fullerton, California
  - Scripps Clinic Green Hospital, La Jolla, California
  - Veterans Administration Hospital, Los Angeles, California
  - University Cardiovascular Medical Group, Los Angeles, California
  - Cardio-Pulmonary Associates, Monterey, California
  - Temecula Valley Cardiology, Murrieta, California
  - California Pacific Cardiovascular Medical, San Francisco, California
  - East Bay Cardiology, San Pablo, California
  - Cardiology Consultants Medical Group, Tarzana, California
  - Medical Center of the Rockies, Fort Collins, Colorado
  - Connecticut Heart & Vascular Center, Bridgeport, Connecticut
  - Cardiology Consultants, PA, Newark, Delaware
  - Heart and Vascular Center of Bradenton, Bradenton, Florida
  - Clearwater Cardiovascular & Intervention, Clearwater, Florida
  - Mahesh Amin, MD PA, Clearwater, Florida
  - Pasco Cardiology, Hudson, Florida
  - Cardiovascular Associates, Kissimmee, Florida
  - Clark and Daughtrey Medical Group, Lakeland, Florida
  - OMNI, Melbourne, Florida
  - Miami Cardiology Group, Miami, Florida
  - Florida Heart Group, Orlando, Florida
  - Cardiology Associates, Port Charlotte, Florida
  - Cardiovascular Consultants,, Tamarac, Florida
  - Indian River Cardiovascular Associate, Vero Beach, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Cardiology of Atlanta, Atlanta, Georgia
  - Northside Cardiology, Atlanta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Southcoast Cardiology, Savannah, Georgia
  - Pacific Cardiology, Honolulu, Hawaii
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - Heart Care Center of Illinois, Blue Island, Illinois
  - MidAmerica Cardiovascular Consultants, Frankfort, Illinois
  - Cardiovascular Associates of Glenbrook and Evanston, LLC, Glenview, Illinois
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - St. Vincent's Hospital Indianapolis, Indianapolis, Indiana
  - St. Vincent's Hospital,, Indianapolis, Indiana
  - Iowa Heart Center PC,, West Des Moines, Iowa
  - Mid America Cardiology, Kansas City, Kansas
  - Cardiology Consultants, Topeka, Kansas
  - Cardiovascular Consultants of Kansas, Wichita, Kansas
  - Louisville Cardiology Medical Group P.S, Louisville, Kentucky
  - Medical Center Cardiologists P.S.C, Louisville, Kentucky
  - Owensboro Heart and Vascular, Owensboro, Kentucky
  - Tchefuncte Cardiovascular Associates,, Covington, Louisiana
  - Heart Clinic of Louisiana, Marrero, Louisiana
  - Maryland Heart, PC, Bethesda, Maryland
  - Heart Center of Southern Maryland, Clinton, Maryland
  - Arundel Heart Associates, Glen Burnie, Maryland
  - Peninsula Cardiology, Salisbury, Maryland
  - Primary Care Specialists Inc, Ayer, Massachusetts
  - Merrimack Valley Cardiology, Chelmsford, Massachusetts
  - Harbor Medical AssociatesSo Weymouth, Weymouth, Massachusetts
  - Consultants in Cardiology, Farmington Hills, Michigan
  - Cardiovascular Consultants PC, Rochester, Michigan
  - Eastside Cardiology, Roseville, Roseville, Michigan
  - St. Paul Cardiology, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - University Hospital Healthcare, Columbia, Missouri
  - Freeman Heart Institute, Joplin, Missouri
  - Mercy Cardiology, St Louis, Missouri
  - Cardiology Diagnostics, Ltd,, St Louis, Missouri
  - Cardiac Associates of New Hampshire, Concord, New Hampshire
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Medicor, Bridgewater, New Jersey
  - Cross County Cardiology, Edgewater, New Jersey
  - Heart-Lung Center, Hawthorne, New Jersey
  - Southern New Jersey Cardiac Specialists, Voorhees Township, New Jersey
  - Diagnostic and Clinical Cardiologists, West Orange, New Jersey
  - Westwood Cardiology, Westwood, New Jersey
  - Albany Associates in Cardiology,, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Cardiology Associates of Brooklyn, Brooklyn, New York
  - United Medical Associates, Brooklyn, New York
  - Concorde Medical Group/NYU Hospital, Manhattan, New York
  - Island Cardiac Specialists, Mineola, New York
  - Island Cardiac Specialist, Mineola, New York
  - Gotham Cardiovascular Research, New York, New York
  - Westchester Medical Group, Scarsdale, New York
  - Vazzana and Bogin Cardiology Associates, Staten Island, New York
  - Cardiology PC, Syracuse, New York
  - Southbay Cardiology, West Islip, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Sanger Clinic, Charlotte, North Carolina
  - Carolina Heart Specialists, Gastonia, North Carolina
  - Southeastern Heart and Vascular, Greensboro, North Carolina
  - Hickory Cardiology, Hickory, North Carolina
  - Carolina Cardiology Associates, High Point, North Carolina
  - Heart Center of Eastern Carolina,, New Bern, North Carolina
  - Heart Center of Eastern Carolina, New Bern, North Carolina
  - Pinehurst Cardiology Consultants, Pinehurst, North Carolina
  - Raleigh Cardiology, Raleigh, North Carolina
  - Meritcare Medical Center, Fargo, North Dakota
  - Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - Muhammed H. Zahra, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Doctors Hospital Heart Failure Clinic, Columbus, Ohio
  - Schuster Cardiology Associates, Kettering, Ohio
  - The Heart Institute of Northwest Ohio, Lima, Ohio
  - Bryce Morrice MD and Debra Heldman MD Inc, Newark, Ohio
  - Cardiovascular Clinic, Inc., Parma, Ohio
  - North West Ohio Cardiology Consultants, Toledo, Ohio
  - Abington Medical Specialists, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Central Bucks Specialists, Ltd.,, Doylestown, Pennsylvania
  - Associated Cardiologists, Harrisburg, Pennsylvania
  - The Heart Group, Ltd, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Cardiology Associates of Southeastern PA, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Blackstone Cardiology Associates, Pawtucket, Rhode Island
  - Medical University of South, Charleston, South Carolina
  - Upstate Cardiology, Greenville, South Carolina
  - Cardiology Associates, Myrtle Beach, South Carolina
  - Cardiology Consultants, PA, Spartanburg, South Carolina
  - Sumter Medical Consultants, Sumter, South Carolina
  - Columbia Cardiology Consultants, West Columbia, South Carolina
  - Sutherland Clinic, Germantown, Tennessee
  - Dela Clinic, Lexington, Tennessee
  - Heart Place North Arlington, Arlington, Texas
  - University of Texas South Western Medical Center at Dallas, Dallas, Texas
  - Comprehensive Heart Care, PA, Houston, Texas
  - Cardiology Consultants of Houston, Houston, Texas
  - Legacy Heart Center, Plano, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - Wilford Hall Medical Center, San Antonio, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - University Associates in Cardiology, Burlington, Vermont
  - Cardiology Associates of Lakeview, Fairfax, Virginia
  - The Cardiovascular Group, Fairfax, Virginia
  - Tidewater Heart Specialists, Inc.,, Hampton, Virginia
  - Cardiology Associates of Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Derived] Shukla A, Curtis AB, Mehra MR, Albert NM, Gheorghiade M, Heywood JT, Liu Y, O'Connor CM, Reynolds D, Walsh MN, Yancy CW, Fonarow GC. Factors associated with improvement in utilization of cardiac resynchronization therapy in eligible heart failure patients: findings from IMPROVE HF. Pacing Clin Electrophysiol. 2013 Apr;36(4):433-43. doi: 10.1111/pace.12090. Epub 2013 Feb 4. PMID 23380000
- [Derived] Barkoudah E, Skali H, Uno H, Solomon SD, Pfeffer MA. Mortality rates in trials of subjects with type 2 diabetes. J Am Heart Assoc. 2012 Feb;1(1):8-15. doi: 10.1161/JAHA.111.000059. Epub 2012 Feb 20. PMID 23130114
- [Derived] Reynolds D, Albert NM, Curtis AB, Gheorghiade M, Heywood JT, Mcbride ML, Inge PJ, Mehra MR, O'Connor CM, Walsh MN, Yancy CW, Fonarow GC. Race and improvements in the use of guideline-recommended therapies for patients with heart failure: findings from IMPROVE HF. J Natl Med Assoc. 2012 May-Jun;104(5-6):287-98. doi: 10.1016/s0027-9684(15)30156-5. PMID 22973678
- [Derived] Fonarow GC, Albert NM, Curtis AB, Gheorghiade M, Heywood JT, Liu Y, Mehra MR, O'Connor CM, Reynolds D, Walsh MN, Yancy CW. Associations between outpatient heart failure process-of-care measures and mortality. Circulation. 2011 Apr 19;123(15):1601-10. doi: 10.1161/CIRCULATIONAHA.110.989632. Epub 2011 Apr 4. PMID 21464053
- [Derived] Walsh MN, Yancy CW, Albert NM, Curtis AB, Gheorghiade M, Heywood JT, Inge PJ, McBride ML, Mehra MR, O'Connor CM, Reynolds D, Fonarow GC. Equitable improvement for women and men in the use of guideline-recommended therapies for heart failure: findings from IMPROVE HF. J Card Fail. 2010 Dec;16(12):940-9. doi: 10.1016/j.cardfail.2010.07.250. PMID 21111983
- [Derived] Fonarow GC, Albert NM, Curtis AB, Stough WG, Gheorghiade M, Heywood JT, McBride ML, Inge PJ, Mehra MR, O'Connor CM, Reynolds D, Walsh MN, Yancy CW. Improving evidence-based care for heart failure in outpatient cardiology practices: primary results of the Registry to Improve the Use of Evidence-Based Heart Failure Therapies in the Outpatient Setting (IMPROVE HF). Circulation. 2010 Aug 10;122(6):585-96. doi: 10.1161/CIRCULATIONAHA.109.934471. Epub 2010 Jul 26. PMID 20660805
- [Derived] Heywood JT, Fonarow GC, Yancy CW, Albert NM, Curtis AB, Gheorghiade M, Inge PJ, McBride ML, Mehra MR, O'Connor CM, Reynolds D, Walsh MN. Comparison of medical therapy dosing in outpatients cared for in cardiology practices with heart failure and reduced ejection fraction with and without device therapy: report from IMPROVE HF. Circ Heart Fail. 2010 Sep;3(5):596-605. doi: 10.1161/CIRCHEARTFAILURE.109.912683. Epub 2010 Jul 15. PMID 20634483
- [Derived] Walsh MN, Yancy CW, Albert NM, Curtis AB, Stough WG, Gheorghiade M, Heywood JT, McBride ML, Mehra MR, O'Connor CM, Reynolds D, Fonarow GC. Electronic health records and quality of care for heart failure. Am Heart J. 2010 Apr;159(4):635-642.e1. doi: 10.1016/j.ahj.2010.01.006. PMID 20362723
- [Derived] Mehra MR, Yancy CW, Albert NM, Curtis AB, Stough WG, Gheorghiade M, Heywood JT, McBride ML, O'Connor CM, Reynolds D, Walsh MN, Fonarow GC. Evidence of clinical practice heterogeneity in the use of implantable cardioverter-defibrillators in heart failure and post-myocardial infarction left ventricular dysfunction: Findings from IMPROVE HF. Heart Rhythm. 2009 Dec;6(12):1727-34. doi: 10.1016/j.hrthm.2009.08.022. Epub 2009 Aug 22. PMID 19959119
- [Derived] Curtis AB, Yancy CW, Albert NM, Stough WG, Gheorghiade M, Heywood JT, McBride ML, Mehra MR, Oconnor CM, Reynolds D, Walsh MN, Fonarow GC. Cardiac resynchronization therapy utilization for heart failure: findings from IMPROVE HF. Am Heart J. 2009 Dec;158(6):956-64. doi: 10.1016/j.ahj.2009.10.011. PMID 19958862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study sites included outpatient cardiology practices in the United States. Patients diagnosed with heart failure or prior myocardial infarction or developed moderate-severe left ventricular dysfunction were included. Each cardiology practice had five chart reviews and an educational workshop as a part of the process improvement intervention.
Pre-assignment Details: The study included 3 mutually exclusive patient cohorts. Patients in cohort A were reviewed at baseline, 12 and 24 months. This is also called the longitudinal cohort. Patients in cohort B and C were reviewed at 6 and 18 months, respectively. These two cohorts are referred to as the single time point cohorts.
Groups:
- Cohort A (Baseline, 12 and 24 Months): Cohort A: The charts of 15,177 patients were reviewed at baseline, 12 months and 24 months. The principal investigator and HF nurse of the study sites attended an educational workshop at baseline, 12 and 24 months as well where they were provided with tools meant to improve HF care at their practices. The tools included tip cards, worksheets, and patient education materials. Cohort A is a longitudinal cohort.
- Cohort B (6 Months): Cohort B: The charts of 9,992 patients were reviewed at 6 months. The principal investigator and HF nurse of the study sites attended an educational workshop at the same time where they were provided with tools meant to improve HF care at their practices. The tools included tip cards, worksheets, and patient education materials. Cohort B is a single time point cohort.
- Cohort C (18 Months): Cohort C: The charts of 9,641 patients were reviewed at 18 months. The principal investigator and HF nurse of the study sites attended an educational workshop at the same time where they were provided with tools meant to improve HF care at their practices. The tools included tip cards, worksheets, and patient education materials. Cohort C is a single time point cohort.
Period: Overall Study
Arm/Group | Cohort A (Baseline, 12 and 24 Months) | Cohort B (6 Months) | Cohort C (18 Months)
Started | 15177 (at baseline) | 9992 (at 6 months) | 9641 (at 18 months)
Completed | 7605 (at 24 Months) | 9992 (at 6 months) | 9641 (at 18 months)
Not Completed | 7572 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Baseline, 12 and 24 Months) | Cohort B (6 Months) | Cohort C (18 Months) | Total
Number analyzed (Participants) | 15177 | 9992 | 9641 | 34810
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (13.2) | 68.3 (13.2) | 68.2 (13.6) | 68.4 (13.3)
Age, Customized [Number; unit: participants]
  <=64 years | 5274 | 3606 | 3539 | 12419
  Between 64 and 76 years | 5127 | 3344 | 3089 | 11560
  >76 years | 4748 | 3041 | 3010 | 10799
  Missing | 28 | 1 | 3 | 32
Sex/Gender, Customized [Number; unit: participants]
  Female | 4383 | 2918 | 2827 | 10128
  Male | 10787 | 7069 | 6814 | 24670
  Missing | 7 | 5 | 0 | 12
Region of Enrollment [Number; unit: participants]
  United States | 15177 | 9992 | 9641 | 34810

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Over the Aggregate IMPROVE-HF Practice Sites the Relative Changes in 7 Performance Measures at 24 Months Compared With Baseline and Determine the Number of Performance Measures That Achieved a Relative 20% or Greater Positive Change.
Description: 7 performance measures: angiotensin converting enzyme inhibitor and/or angiotensin II receptor blockers (ACEI/ARB), beta-blokers, aldosterone receptor antagonists, anticoagulation for atrial fibrillation (AF), cardiac resynchronization therapy (CRT-P/CRT-D), cardioverter-defibrillator (ICD/CRT-D), heart failure (HF) education.
  We first calcuated % of patients who were eligible for a performance measure that were treated by it at baseline and 24 months. We then calculated the relative change as (% treated at 24 months - % treated at baseline)/% treated at baseline. The 95% confidence interval (CI) was calculated and the relative change of each performance measure was evaluated using a z-test for one-sample proportion.
  The number of performance measures with >= 20% relative improvement was determined. The intervention was considered successful if a relative 20% or greater improvement in at least 2 of the 7 performance measures at 24 months compared with baseline was achieved.
Time Frame: 24 Month
Population: 167 practices contributed data to the baseline chart review. Twelve of the practices withdrew from the study prior to the next chart review milestone. 155 of those practices' data contributed to the follow up of the longitudinal cohort time points of 12 and 24 months post educational workshop.
Measure: Number (95% Confidence Interval); unit: percentage of participants in aggregate
Groups:
- Cohort A (at Baseline): For this longitudinal cohort, data are collected at baseline, 12 months and 24 months after the principle investigator and HF nurse attend an educational workshop. All longitudinal analyses will be performed on this cohort of patients. This arm includes all the atients at baseline. Percentage of patients who were eligible for a performance measure that were treated by it at baseline was calculated.
- Cohort A (at 24 Months): For this longitudinal cohort, data are collected at baseline, 12 months and 24 months after the principle investigator and HF nurse attend an educational workshop. All longitudinal analyses will be performed on this cohort of patients. This arm includes the completers, i.e. patients who have a qualifying visit at both baseline and 24 months who were living at the 24 month chart review and are qualified for at least one performance measure at 24 months. Percentage of the patients who were eligible for a performance measure that were treated by it at the 24 months was calculated.
- Cohort A (Relative Change 24 Months vs. Baseline): For this longitudinal cohort, data are collected at baseline, 12 months and 24 months after the principle investigator and HF nurse attend an educational workshop. All longitudinal analyses will be performed on this cohort of patients. This arm includes the completers, i.e. patients who have a qualifying visit at both baseline and 24 months who were living at the 24 month chart review and are qualified for at least one performance measure at 24 months. The relative changes in the percentages from 24 months to baseline were calculated for the 7 performance measures.
Arm/Group | Cohort A (at Baseline) | Cohort A (at 24 Months) | Cohort A (Relative Change 24 Months vs. Baseline)
Number analyzed (Participants) | 15177 | 7605 | 7605
percentage of participants in aggregate
  Performance Measure 1: ACEI/ARB | 79.8 [79.2 to 80.5] | 86.5 [85.6 to 87.3] | 8.4 [7.0 to 9.7]
  Performance Measure 2: Beta-blocker | 86.2 [85.6 to 86.8] | 93.6 [93.0 to 94.2] | 8.6 [7.7 to 9.6]
  Performance Measure 3: Aldosterone antagonist | 34.4 [32.7 to 36.1] | 61.8 [59.2 to 64.5] | 79.7 [70.5 to 89.0]
  Performance Measure 4: Anticoagulation for AF | 68.6 [67.2 to 70.0] | 69.3 [67.5 to 71.0] | 1.0 [-2.2 to 4.2]
  Performance Measure 5: CRT-P/CRT-D | 37.7 [35.2 to 40.1] | 68.5 [65.8 to 71.3] | 81.9 [72.2 to 91.7]
  Performance Measure 6: ICD/CRT-D | 48.8 [47.8 to 49.8] | 79.1 [78.0 to 80.2] | 62.1 [59.1 to 65.1]
  Performance Measure 7: HF education | 61.8 [61.0 to 62.5] | 70.8 [69.8 to 71.9] | 14.7 [12.6 to 16.8]
Statistical Analysis 1: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #1: relative change in % of eligible patients treated with angiotensin converting enzyme inhibitor and/or angiotensin II receptor blockers (ACEU/ARB); Test type: Superiority or Other; p < 0.001, a large sample test (z-test); Relative Improvement (%) = 8.4, 95% CI 2-sided [7.0 to 9.7]
Statistical Analysis 2: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #2: relative change in % of eligible patients treated with beta-blockers; Test type: Superiority or Other; p < 0.001, a large sample test (z-test); Relative improvement (%) = 8.6, 95% CI 2-sided [7.7 to 9.6]
Statistical Analysis 3: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #3: relative change in % of eligible patients treated with aldosterone receptor antagonists; Test type: Superiority or Other; p < 0.001, a large sample test (z-test); Relative improvement (%) = 79.7, 95% CI 2-sided [70.5 to 89.0]
Statistical Analysis 4: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #4: relative change in % of eligible patients treated with anticoagulation for AF; Test type: Superiority or Other; p = 0.546, a large sample test (z-test); Relative Improvement (%) = 1.0, 95% CI 2-sided [-2.2 to 4.2]
Statistical Analysis 5: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #5: relative change in % of eligible patients treated with cardiac resynchronization therapy (CRT-P/CRT-D); Test type: Superiority or Other; p < 0.001, a large sample test (z-test); Relative Improvement (%) = 81.9, 95% CI 2-sided [72.2 to 91.7]
Statistical Analysis 6: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #6: relative change in % of eligible patients treated with implantable cardioverter-defibrillator (ICD) or CRT-D; Test type: Superiority or Other; p < 0.001, a large sample test (z-test); Relative Improvement (%) = 62.1, 95% CI 2-sided [59.1 to 65.1]
Statistical Analysis 7: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #7: relative change in % of eligible patients with HF education; Test type: Superiority or Other; p < 0.001, a large sample test (z-test); Relative Improvement (%) = 14.7, 95% CI 2-sided [12.6 to 16.8]

2. Secondary Outcome: Observe the Number of Sites That Demonstrate a Relative 20% or Greater Improvement in 2 or More of the 7 Performance Measures at 24 Months as Compared to Baseline in Cohort A.
Description: The number of practices that achieved greater than or equal to 20% improvement in two or more of the 7 performance measures at 24 months as compared to baseline of cohort A is presented.
Time Frame: 24 months
Measure: Number; unit: Sites
Units Other Than Participants: Sites
Groups:
- Practice Sites in Cohort A: In this analysis, 167 practices contributed data to the baseline chart review of Cohort A. Of them, 12 practices withdrew from the study prior to the next chart review milestone. Therefore, 155 practices' data contributed to the follow up of the longitudinal cohort time points of 12 and 24 months post educational workshop. Correspondingly there were 7605 patients whose chart review was completed at both baseline and 24 months.
Arm/Group | Practice Sites in Cohort A
Number analyzed (Participants) | 7605
Number analyzed (Sites) | 155
Sites
  Performance Measure 1: ACEI/ARB | 15
  Performance Measure 2: Beta-blocker | 9
  Performance Measure 3: Aldosterone antagonist | 82
  Performance Measure 4: Anticoagulation for AF | 14
  Performance Measure 5: CRT-P/CRT-D | 83
  Performance Measure 6: ICD/CRT-D | 114
  Performance Measure 7: HF education | 59
  >=20% relative change in 2 or more measures | 123

3. Secondary Outcome: Observe the Change From Baseline to 24 Months in Each Performance Measure and Composite Score for the Aggregate Practices.
Description: performance measure improvement for each performance measure was analyzed at a practice level from baseline to 24 months. Performance measure adherence was calculated at the individual practice level and then combined and summarized. Mean, standard deviation, and 95% confidence intervals for performance measure adherence, composite score and relative change (24 months compared with baseline) are reported.
  The Composite Score is based on the ratio of the sum of the numerators of all individual performance measures to the sum of the denominators of all individual performances measures. The numerator of a performance measure is the number of patients treated with that measure. The denomiator of a performance measure is the number of patients eligible for being treated with that measure.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: Sites
Groups:
- Cohort A (at Baseline): Cohort A at baseline included 15177 patients from 167 study sites (practices).
- Cohort A (at 24 Months): Cohort A at 24 months included 7605 patients from 155 study sites (practices).
- Cohort A (Relative Change 24 Months vs. Baseline): The ralative changes in performance measures and compsite score at 24 months compared to baseline were calculated based on 155 study sites that involved 7605 patients.
Arm/Group | Cohort A (at Baseline) | Cohort A (at 24 Months) | Cohort A (Relative Change 24 Months vs. Baseline)
Number analyzed (Participants) | 15177 | 7605 | 7605
Number analyzed (Sites) | 167 | 155 | 155
percentage
  Performance Measure 1: ACEI/ARB | 78.3 (11.5) | 85.1 (10.6) | 19.4 (128.9)
  Performance Measure 2: Beta-blocker | 86.0 (10.8) | 92.2 (9.8) | 7.6 (16.1)
  Performance Measure 3: Aldosterone antagonist | 34.5 (18.5) | 60.3 (25.9) | 30.0 (33.8)
  Performance Measure 4: Anticoagulation for AF | 68.0 (16.1) | 67.8 (18.0) | 1.0 (28.5)
  Performance Measure 5: CRT-P/CRT-D | 37.2 (30.5) | 66.3 (29.0) | 48.4 (62.3)
  Performance Measure 6: ICD/CRT-D | 50.1 (17.5) | 77.5 (16.8) | 70.9 (62.4)
  Performance Measure 7: HF education | 59.5 (23.7) | 72.1 (24.0) | 50.6 (147.7)
  Composite Score | 67.1 (8.9) | 79.0 (9.3) | 19.2 (18.1)
Statistical Analysis 1: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #1: Relative change at 24 months compared with baseline in ACEI/ARB for the aggregate practices; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; Mean Relative Change (%) = 19.4, 95% CI 2-sided [-1.1 to 39.8]
Statistical Analysis 2: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #2: the relative change at 24 months compared with baseline in beta-blockers for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 7.6, 95% CI 2-sided [5.1 to 10.2]
Statistical Analysis 3: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #3: the relative change at 24 months compared with baseline in aldosterone antagonist for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 30.0, 95% CI 2-sided [24.6 to 35.5]
Statistical Analysis 4: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #4: the relative change at 24 months compared with baseline in anticoagulation for AF for the aggregate practices; Test type: Superiority or Other; p = 0.513, t-test, 2 sided; Mean Relative Change (%) = 1.0, 95% CI [-3.6 to 5.5]
Statistical Analysis 5: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #5: the relative change at 24 months compared with baseline in CRT-P/CRT-D for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 48.4, 95% CI 2-sided [37.9 to 58.8]
Statistical Analysis 6: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #6: the relative change at 24 months compared with baseline in ICD/CRT-D for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 70.9, 95% CI 2-sided [61.0 to 80.8]
Statistical Analysis 7: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Performance Measure #7: the relative change at 24 months compared with baseline in HF education for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 50.6, 95% CI 2-sided [27.1 to 74.2]
Statistical Analysis 8: Comparison: Cohort A (Relative Change 24 Months vs. Baseline); Composite Score: The relative change at 24 months compared with baseline in composite score for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 19.2, 95% CI 2-sided [16.3 to 22.0]

4. Secondary Outcome: Observe the Relative Change Between Baseline of Cohort A and 6 Months of Cohort B in Performance Measures and Composite Score for the Aggregate Practices.
Description: The relative changes between baseline of cohort A and 6 months of cohort B in performance measures and composite score for the aggregate practices were calculated using mean, standard deviation and 95% CI.
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: percentage of participants
Units Other Than Participants: Sites
Groups:
- Cohort A: Baseline: In this analysis, data of Cohort A at baseline were used. This included 15177 patients from 167 cardiology practices.
- Cohort B: 6 Months: In this analysis, data of Cohort B (i.e. 6 months single time point cohort) were used. This included 9992 patients from 154 cardiology practices.
- Cohort B 6 Months vs. Cohort A Baseline (Relative Change): The relative changes in performance measures and composite score of Cohort B (6 months) compared with those of Cohort A at baseline were calculated
Arm/Group | Cohort A: Baseline | Cohort B: 6 Months | Cohort B 6 Months vs. Cohort A Baseline (Relative Change)
Number analyzed (Participants) | 15177 | 9992 | 25169
Number analyzed (Sites) | 167 | 154 | 167
percentage of participants
  Performance Measure 1: ACEI/ARB | 78.7 (11.3) | 80.2 (10.6) | 10.3 (97.1)
  Performance Measure 2: Beta-blocker | 85.9 (10.9) | 90.0 (7.2) | 10.6 (68.9)
  Performance Measure 3: Aldosterone antagonist | 34.7 (18.7) | 33.4 (20.7) | -1.1 (27.4)
  Performance Measure 4: Anticoagulation for AF | 67.9 (15.8) | 68.9 (17.4) | 6.2 (38.2)
  Performance Measure 5: CRT-P/CRT-D | 37.6 (30.7) | 34.9 (27.8) | -1.8 (53.7)
  Performance Measure 6: ICD/CRT-D | 49.9 (17.0) | 52.7 (17.4) | 14.4 (46.9)
  Performance Measure 7: HF education | 59.4 (23.6) | 67.5 (20.8) | 38.5 (94.8)
  Composite Score | 67.1 (8.8) | 70.7 (8.0) | 6.6 (15.1)
Statistical Analysis 1: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Performance Measure #1: the relative change of Cohort B (6 months) compared with Cohort A at baseline in ACEI/ARB for the aggregate practices; Test type: Superiority or Other; p = 0.197, t-test, 2 sided; Mean Relative Change (%) = 10.3, 95% CI 2-sided [-5.4 to 25.9]
Statistical Analysis 2: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Performance Measure #2: the relative change of Cohort B (6 months) compared with Cohort A at baseline in beta-blockers for the aggregate practices; Test type: Superiority or Other; p = 0.061, t-test, 2 sided; Mean Relative Change (%) = 10.6, 95% CI 2-sided [-0.5 to 21.7]
Statistical Analysis 3: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Performance Measure #3: the relative change of Cohort B (6 months) compared with Cohort A at baseline in aldosterone antagonist for the aggregate practices; Test type: Superiority or Other; p = 0.622, t-test, 2 sided; Mean Relative Change (%) = -1.1, 95% CI 2-sided [-5.7 to 3.4]
Statistical Analysis 4: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Performance Measure #4: the relative change of Cohort B (6 months) compared with Cohort A at baseline in anticoagulation for AF for the aggregate practices; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Relative Change (%) = 6.2, 95% CI 2-sided [0.0 to 12.4]
Statistical Analysis 5: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Performance Measure #5: the relative change of Cohort B (6 months) compared with Cohort A at baseline in CRT-P/CRT-D for the aggregate practices; Test type: Superiority or Other; p = 0.711, t-test, 2 sided; Mean Relative Change (%) = -1.8, 95% CI 2-sided [-11.2 to 7.7]
Statistical Analysis 6: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Performance Measure #6: the relative change of Cohort B (6 months) compared with Cohort A at baseline in ICD/CRT-D for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 14.4, 95% CI 2-sided [6.9 to 22.0]
Statistical Analysis 7: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Performance Measure #7: the relative change of Cohort B (6 months) compared with Cohort A at baseline in HF education for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 38.5, 95% CI 2-sided [23.2 to 53.8]
Statistical Analysis 8: Comparison: Cohort B 6 Months vs. Cohort A Baseline (Relative Change); Composite Score: the relative change of Cohort B (6 months) compared with Cohort A at baseline in composite score for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 6.6, 95% CI 2-sided [4.2 to 9.0]

5. Secondary Outcome: Observe the Relative Change Between Baseline of Cohort A and 18 Months of Cohort C in Performance Measures and Composite Score for the Aggregate Practices.
Description: The relative changes between baseline of cohort A and 18 months of cohort C in performance measures and composite score for the aggregate practices were calculated using mean, standard deviation and 95% CI.
Time Frame: baseline and 18 Months
Measure: Mean (Standard Deviation); unit: percentage of participants
Units Other Than Participants: Sites
Groups:
- Cohort C (18 Months): In this analysis, data of Cohort C (i.e. 18 months single time point cohort) were used. This included 9641 patients from 150 cardiology practices.
- Cohort C 18 Months vs. Cohort A Baseline (Relative Change): The relative changes in performance measures and composite score of Cohort C (18 months) compared with those of Cohort A at baseline were calculated.
Arm/Group | Cohort A: Baseline | Cohort C (18 Months) | Cohort C 18 Months vs. Cohort A Baseline (Relative Change)
Number analyzed (Participants) | 15177 | 9641 | 24818
Number analyzed (Sites) | 167 | 150 | 167
percentage of participants
  Performance Measure 1: ACEI/ARB | 78.7 (11.3) | 80.3 (12.2) | 10.5 (97.9)
  Performance Measure 2: Beta-blocker | 85.9 (10.9) | 91.8 (7.0) | 14.3 (87.7)
  Performance Measure 3: Aldosterone antagonist | 34.7 (18.7) | 36.6 (23.1) | 5.8 (58.3)
  Performance Measure 4: Anticoagulation for AF | 67.9 (15.8) | 69.6 (17.1) | 6.7 (38.3)
  Performance Measure 5: CRT-P/CRT-D | 37.6 (30.7) | 43.5 (30.1) | 9.3 (59.7)
  Performance Measure 6: ICD/CRT-D | 49.9 (17.0) | 54.0 (17.2) | 17.6 (51.3)
  Performance Measure 7: HF education | 59.4 (23.6) | 75.0 (22.6) | 59.5 (158.5)
  Composite Score | 67.1 (8.8) | 73.2 (8.4) | 10.6 (18.5)
Statistical Analysis 1: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Performance Measure #1: the relative change of Cohort C (18 months) compared with Cohort A at baseline in ACEI/ARB for the aggregate practices; Test type: Superiority or Other; p = 0.190, t-test, 2 sided; Mean Relative Change (%) = 10.5, 95% CI 2-sided [-5.3 to 26.3]
Statistical Analysis 2: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Performance Measure #2: the relative change of Cohort C (18 months) compared with Cohort A at baseline in beta-blockers for the aggregate practices; Test type: Superiority or Other; p = 0.048, t-test, 2 sided; Mean Relative Change (%) = 14.3, 95% CI 2-sided [0.1 to 28.4]
Statistical Analysis 3: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Performance Measure #3: the relative change of Cohort C (18 months) compared with Cohort A at baseline in aldosterone antagonist for the aggregate practices; Test type: Superiority or Other; p = 0.240, t-test, 2 sided; Mean Relative Change (%) = 5.8, 95% CI 2-sided [-3.9 to 15.4]
Statistical Analysis 4: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Performance Measure #4: the relative change of Cohort C (18 months) compared with Cohort A at baseline in anticoagulation for AF for the aggregate practices; Test type: Superiority or Other; p = 0.033, t-test, 2 sided; Mean Relative Change (%) = 6.7, 95% CI 2-sided [0.5 to 13.0]
Statistical Analysis 5: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Performance Measure #5: the relative change of Cohort C (18 months) compared with Cohort A at baseline in CRT-P/CRT-D for the aggregate practices; Test type: Superiority or Other; p = 0.085, t-test, 2 sided; Mean Relative Change (%) = 9.3, 95% CI 2-sided [-1.3 to 19.8]
Statistical Analysis 6: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Performance Measure #6: the relative change of Cohort C (18 months) compared with Cohort A at baseline in ICD/CRT-D for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 17.6, 95% CI 2-sided [9.3 to 25.8]
Statistical Analysis 7: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Performance Measure #7: the relative change of Cohort C (18 months) compared with Cohort A at baseline in HF education for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 59.5, 95% CI 2-sided [33.9 to 85.2]
Statistical Analysis 8: Comparison: Cohort C 18 Months vs. Cohort A Baseline (Relative Change); Composite Score: the relative change of Cohort C (18 months) compared with Cohort A at baseline in composite score for the aggregate practices; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Relative Change (%) = 10.6, 95% CI 2-sided [7.6 to 13.6]

ADVERSE EVENTS:
Description: Adverse events were not collected for this study.
Arm/Group | Cohort A (Baseline, 12 and 24 Months) | Cohort B (6 Months) | Cohort C (18 Months)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigation Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication. PI's may not publish single-site data until the main multi-site publication has occurred.